CLINICAL TRIAL: NCT02519621
Title: A Pilot Study to Compare the Efficacy of NPWT PRO Versus KCI Ulta® NPWT and to Compare NPWT PRO Versus NPWT PRO With Simultaneous Irrigation on Wound Healing
Brief Title: NPWT PRO vs KCI Ulta® NPWT and to Compare NPWT PRO vs NPWT PRO With Simultaneous Irrigation on Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larry Lavery (Other)
Responsible Party: Sponsor-Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 032015-099
Record Dates: First submitted 2015-06-01; First posted 2015-08-11 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Partial-thickness Burn; Ulcer
Keywords: diabetic ulcer; pressure ulcer; chronic or traumatic wound; sub-acute or dehisced wound
MeSH Terms: conditions — Ulcer; Pressure Ulcer; Bronchiolitis Obliterans Syndrome | interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NPWT PRO without irrigation (Active Comparator): Cardinal Health NPWT PRO system (K143016) continuous/intermittent vacuum-assisted drainage
  Interventions: Device: NPWT PRO without irrigation
- NPWT PRO with Irrigation (Active Comparator): Cardinal Health NPWT PRO system (K143016) continuous/intermittent vacuum-assisted drainage with simultaneous delivery of topical wound treatment solutions and suspensions over the wound bed (saline irrigant).
  Interventions: Device: NPWT PRO with irrigation
- KCI Ulta NPWT (Active Comparator): KCI Ulta NPWT without irrigation.
  Interventions: Device: KCI Ulta

INTERVENTIONS:
Device: NPWT PRO without irrigation — NPWT PRO without irrigation.
  Other Names: Cardinal Quantum NPWT PRO
  Arms: NPWT PRO without irrigation
Device: NPWT PRO with irrigation — NPWT PRO with irrigation (saline)
  Other Names: Cardinal Quantum NPWT PRO
  Arms: NPWT PRO with Irrigation
Device: KCI Ulta — KCI Ulta NPWT without irrigation
  Arms: KCI Ulta NPWT

SUMMARY:
This study is designed to assess the efficacy and economics of two NPWT (negative pressure wound therapy) branded devices of wound healing outcomes. It is also designed to assess the effectiveness of negative pressure and negative pressure with continuous irrigation on multiple parameters of wound healing. It is a single-center, open-label, active controlled, parallel-group trial that aims to determine the efficacy of Quantum with simultaneous irrigation in the treatment of diabetic foot ulcers. Specifically, eligible participants will be randomized to receive either PRO negative press therapy with simultaneous irrigation; or PRO negative pressure therapy without irrigation; or KCI Ulta negative pressure therapy. Outcomes will include rates of wound healing, time to closure, number of surgeries, length of stay, and days to heal.

DETAILED DESCRIPTION:
Subjects will be taken to the operating room for the initial debridement procedure of the wound. At the end of the procedure, subjects who continue to meet all inclusion and no exclusion criteria will be randomized in a 1:1:1 ratio to be treated with either PRO, PRO with simultaneous irrigation (PROI), or KCI Ulta NPWT. Prior to study initiation sealed prenumbered randomization envelopes will be provided to the research staff and used to obtain randomization assignment. Opening of the randomization envelope will occur intraoperatively at the conclusion of the initial surgical debridement of the wound and conformation of all eligibility requirements. Study staff will use the randomization number labels contained in the envelop. The number will become the subject ID. The assignment will be subjects randomized to PRO, PRO with simultaneous irrigation, or KCI Ulta NPWT.

The research staff will note treatment assignments on the intra operative randomization CRF and instruct the investigator. Treatment therapy wound dressings will be applied in the operating room or in the patient's room immediately after surgery per the investigators discretion, according to the manufacturer's recommendations. In order to ensure consistent study treatment, subjects will receive assigned treatment therapies within their study arm after the initial and any subsequent surgical debridements until the wound is deemed ready for closure or coverage by the Investigator. Subjects randomized to the PRO with simultaneous irrigation Treatment arm are the only subjects that will receive irrigation therapy at any time during the study treatment period. If irrigation therapy is discontinued, subjects in the Treatment arm will transition to PRO NPWT without irrigation. Subjects randomized to the PRO Control arm will receive NPWT only from the PRO therapy unit.

ELIGIBILITY:
Inclusion Criteria:

* Presents with an existing chronic or traumatic wound, sub-acute or dehisced wound, partial-thickness burn, ulcer (such as a diabetic or pressure ulcer), flap or graft as diagnosed by a qualified and certified medical practitioner (M.D., D.O., or D.P.M)
* Wound presents with full thickness loss of epidermis and dermis
* The presentation of a wound that in the opinion of the investigators will require surgical debridement, and the wound is expected to be a good candidate for NPWT and eventual wound closure.
* ABI≥0.5 or toe pressures >30 PVR/mmHg
* Subject is willing and able to abstain from partaking in any other form of treatment for his or her wound throughout the duration of his or her course of participation in the clinical study, other than the study procedures described herein.
* 18 years of age or older

Exclusion Criteria:

* Does not present with an existing chronic or traumatic wound, sub-acute or dehisced wound, partial-thickness burn, ulcer (such as a diabetic or pressure ulcer), flap or graft, or a definitive diagnosis cannot be made, as diagnosed by a qualified and certified medical practitioner (M.D., D.O., or D.P.M)
* Wound does not present with full thickness loss of epidermis and dermis
* ABI<0.5 or toe pressures <30 PVR/mmHg
* Subject is not willing or is not able or it is not medically prudent for the subject to abstain from partaking in any other form of treatment for his or her wound throughout the duration of his or her course of participation in the clinical study, other than the study procedures described.
* Subject is unwilling or unable to use the NPWT device at home
* Active Charcot arthropathy
* Collagen vascular disease
* Scleroderma
* Non-enteric and unexplored fistula
* Necrotic tissue with eschar present after debridement
* General skin disorder in the area of the wound such as psoriasis or penicilitis
* Malnutrition (defined as BMI <19)
* Hypercoagulable state based on documentation in their medical record
* Acute deep vein thrombosis
* Current active malignancy in the wound
* Current melanoma or history of melanoma at the wound
* Current active or history of invasive squamous cell carcinoma at the wound
* Sepsis (defined as positive blood culture with leukocytosis) and temperature >101.5 at the time of screening
* Significant Hematologic disorders EXCLUDING anemia
* HIV
* Fever at screening > 101.5
* Deep X-ray therapy
* Untreated bone or soft tissue infection (osteomyelitis)
* Any concomitant illness(es) or medical condition(s) that in the opinion of the investigator would render the subject not suited for study participation
* Subject is taking a regimen of any medication(s) in a significant enough dosage that may affect chronic wound healing, including corticosteroid, chemotherapeutic and non-steroidal anti-inflammatory (NSAID) medications
* Less than 18 years of age
* Developmental disability/significant psychological disorder that could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
* Females currently pregnant or planning pregnancy during the course of intended participation in the study
* Active alcohol or substance abuse in the opinion of the investigator that could impair the subjects ability to provide informed consent, participate in the study protocol or record study measures.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Southwestern, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 93 were consented but 3 of them did not have the vac/treatment, so therefore 90 total (30 in each group).
Period: Overall Study
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.50 (9.95) | 53.80 (12.21) | 51.70 (9.44) | 51.67 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 4 | 16
  Male | 25 | 23 | 26 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10 | 1 | 5 | 16
  African American | 4 | 9 | 1 | 14
  Hispanic | 16 | 20 | 24 | 60
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Complete Wound Healing
Description: Complete healing of wounds as defined by epithelialization with no drainage in three treatment arms: NPWT PRO versus KCI Ulta® NPWT and to Compare NPWT PRO versus NPWT PRO with Simultaneous Irrigation
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT
Number analyzed (Participants) | 30 | 30 | 30
Participants | 15 | 19 | 14

2. Secondary Outcome: Number of Surgeries
Description: Number of surgeries required to debride infection before wound was ready for closure or coverage.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: surgeries
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT
Number analyzed (Participants) | 30 | 30 | 30
surgeries | 2.4 (0.77) | 2.0 (0.49) | 2.4 (0.68)

3. Secondary Outcome: Length of Stay
Description: Number of days the patient stayed in the hospital
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT
Number analyzed (Participants) | 30 | 30 | 30
days | 14.7 (7.4) | 16.3 (15.7) | 15.3 (10.5)

4. Secondary Outcome: Days to Heal
Description: The number of days to heal the wound after last surgery was performed.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT
Number analyzed (Participants) | 30 | 30 | 30
days | 41.0 (6.3) | 43.0 (9.4) | 42.0 (13.1)

ADVERSE EVENTS:
Time Frame: Adverse events during 12 weeks
Arm/Group | NPWT PRO Without Irrigation | NPWT PRO With Irrigation | KCI Ulta NPWT
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 4/30 | 4/30
Other Adverse Events (participants affected / at risk) | 4/30 | 5/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPWT PRO Without Irrigation (N=30) | NPWT PRO With Irrigation (N=30) | KCI Ulta NPWT (N=30)
Foot related readmission (Infections and infestations) | 4 (4) | 4 (4) | 4 (4) — Serious adverse event - readmission to the hospital for foot-related problem.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPWT PRO Without Irrigation (N=30) | NPWT PRO With Irrigation (N=30) | KCI Ulta NPWT (N=30)
Reinfection of study foot (Infections and infestations) | 4 (4) | 5 (5) | 5 (5) — New infection of the study foot during the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02519621/Prot_SAP_000.pdf